CLINICAL TRIAL: NCT03889236
Title: The Effect of Dietary Interventions on Endothelial Glycocalyx Dimensions and Barrier Function in South Asian Patients With Diabetic Nephropathy.
Brief Title: Dietary Interventions on Glycocalyx Dimensions in South Asian Patients With Diabetic Nephropathy.
Acronym: Glycotreat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other); Health Holland (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, AnoukvanderVelden, Msc., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P17.249
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Nephropathy Type 2; Albuminuria; Type2 Diabetes Mellitus; Glucose Metabolism Disorders; Microalbuminuria; Diabetic Nephropathies; Diabetic Complications Renal; Diabetes Mellitus; Kidney Diseases; South Asian
MeSH Terms: conditions — Albuminuria; Glucose Metabolism Disorders; Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — Gestyl

STUDY DESIGN:
Intervention Model Description: Patients are randomized into the diet group, food supplement group or placebo group. The placebo and foodsupplement groups are double blinded.
Who Masked: Participant, Investigator
Masking Description: The placebo and food supplement groups are double blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting mimicking diet (Experimental): 5-day Fasting mimicking diet Prolon. In total 3 cycles of the FMD in three months.
  Interventions: Other: Fasting mimicking diet Prolon
- Food supplement (Experimental): 4 capsules a day of the food supplement Endocalyx for 3 months.
  Interventions: Dietary Supplement: Food supplement Endocalyx
- Placebo (Placebo Comparator): 4 capsules a day of the placebo for 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Other: Fasting mimicking diet Prolon — 5-day fasting mimicking diet
  Other Names: FMD; Prolon; L-Nutra
  Arms: Fasting mimicking diet
Dietary Supplement: Food supplement Endocalyx — Food supplement
  Other Names: Endocalyx; Q-prime
  Arms: Food supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Evaluate the effect of a fasting mimicking diet and a food supplement on the microvascular health and urinary heparanase levels in South Asian type 2 diabetic patients with albuminuria.

ELIGIBILITY:
Inclusion Criteria:

1. South Asian patient with diabetes mellitus type 2.
2. Female or male, aged between 18 and 75 years.
3. Body Mass Index ≥18.5.
4. CKD-EPI >45 ml/min/1.73m² .
5. Proven microalbuminuria defined as albumin/creatinine ratio ≥0.3 and <30 mg/mmol (single portion) or 3-300 mg albumin per day (24 hours urine collection) in the last twelve months.
6. Systolic blood pressure ≤ 180 mmHg.
7. Treatment with hypoglycemic drugs: metformin, sulphonylureas and/or insulin.
8. Subject is willing to participate in the study, must be able to give informed consent and the consent must be obtained prior to any study procedure.
9. Patients must be able to adhere to the study visit schedule and protocol requirements.
10. If female and of child-bearing age, patients must be non-pregnant, non-breastfeeding, and use adequate contraception.

4.3 Exclusion

Exclusion Criteria:

1. Any concurrent illness, disability or clinically significant abnormality that may, as judged by the investigator, affect the interpretation of clinical efficacy or safety data or prevent the subject from safely completing the assessments required by the protocol.
2. Non-diabetic renal disease e.g. known polycystic kidney disease.
3. Use of LMW heparin and/or immunosuppressive drugs.
4. Significant food allergies for galactose, nuts, soy, tomato, corn, grape, melon and artichoke, which would make the subject unable to consume the food provided.
5. Signs of active infection or autoimmune disease, requiring systemic treatment.
6. A psychiatric, addictive or any disorder that compromises ability to give truly informed consent for participation in this study.
7. Malignancy (including lymphoproliferative disease) within the past 2-5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
8. Use of any other investigational drug.
9. Patient has enrolled another clinical trial within last 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in the Microvascular Health Index in the fasting mimicking diet or food supplement group compared to the placebo group | 3 months

SECONDARY OUTCOMES:
Percentage change from baseline in Urine albumin-to-creatinine ratio (UACR) in the fasting mimicking diet or food supplement group compared to the placebo | 3 months
Percentage change from baseline in urinary heparanase levels in the fasting mimicking diet or food supplement group compared to the placebo | 3 months
Percentage change from baseline in urinary MCP-1 levels in the fasting mimicking diet or food supplement group compared to the placebo | 3 months
Percentage change from baseline in specific urinary heparan sulfate domains in the fasting mimicking diet or food supplement group compared to the placebo | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ton J. Rabelink, Prof., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden Universitiy Medical Center (LUMC), Leiden, North Holland, Netherlands

REFERENCES:
- [Derived] van der Velden AIM, IJpelaar DHT, Chandie Shaw PK, Pijl H, Vink H, van der Vlag J, Rabelink TJ, van den Berg BM. Role of dietary interventions on microvascular health in South-Asian Surinamese people with type 2 diabetes in the Netherlands: A randomized controlled trial. Nutr Diabetes. 2024 Apr 10;14(1):17. doi: 10.1038/s41387-024-00275-5. PMID 38600065

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03889236/Prot_SAP_000.pdf